CLINICAL TRIAL: NCT03942952
Title: PEDIATRIC SONICS: Pediatric Study of Neuropsychology and Imaging in CNS Demyelinating Syndromes.
Acronym: SONICS
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Benjamin Greenberg, Professor, University of Texas Southwestern Medical Center
Other Study IDs: STU-2019-0491
Record Dates: First submitted 2019-04-22; First posted 2019-05-08 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting; Neuromyelitis Optica; Acute Disseminated Encephalomyelitis; Transverse Myelitis
Keywords: Multiple Sclerosis; NMO; anti-MOG; Acute Disseminated Encephalolmyelitis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Neuromyelitis Optica; Encephalomyelitis, Acute Disseminated; Myelitis, Transverse; Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CNS demyelinating diagnosis: Diagnosis of CNS demyelinating disorder: Multiple Sclerosis, Transverse Myelitis, Neuromyelitis Optica, Acute Disseminated Encephalomyelitis, anti-MOG antibody, Optic Neuritis.
  * 3T and 7T MRI
  * Neuropsychological testing
  * Optical Coherence Tomography
  * Questionnaires: Quality of Life and Behavior scales
  * Non invasive clinical assessment : Walking, hand and eye coordination tests Repeat same research activities one to year and a half year later
- Healthy Control: * 3T and 7T MRI
  * Neuropsychological testing
  * Optical Coherence Tomography
  * Questionnaires: Quality of Life and Behavior scales
  * Non invasive clinical assessment : Walking, hand and eye coordination tests Repeat same research activities one year to a year and a half later

SUMMARY:
Central Nervous System (CNS) demyelinating conditions include multiple sclerosis (MS), Acute Disseminated Encephalomyelitis (ADEM), Neuromyelitis Optica Spectrum Disorder (NMOSD), Optic Neuritis (ON) and Transverse Myelitis (TM). The symptoms of these conditions are quite variable from patient to patient, but can include motor, sensory, visual, gait and cognitive changes. Conventional MRI can be used to look for new anatomic changes, but fails to measure underlying biochemical changes in brain tissue. The purposes of this study are to identify the biologic and anatomic correlations between cognitive profiles and disease activity using MRI imaging techniques.

DETAILED DESCRIPTION:
Pediatric patients (age 12 to 21 inclusive) with a diagnosis of multiple sclerosis, ADEM, anti-MOG mediated demyelinating disease as well as healthy controls will be recruited to undergo clinical testing. The study visits will include neuropsychological testing, optical coherence tomography (OCT) and MRI on both the 3T and 7T magnet. Subjects will be asked to undergo two study visits separated by 12 months to 18 months. Each study visit will have the same neuropsychological, OCT, and research MRI examinations.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Multiple Sclerosis , ADEM, anti-MOG antibody associated CNS demyelination
2. Age 12 to 21 inclusive at time of enrollment
3. Ability of parent or legal guardian to provide informed consent if participant is under 18.
4. Ability of patients age 12-17 to give assent
5. Completion of the signed HIPPA authorization form by a parent or legal guardian or by participants (18 years of age).

Exclusion Criteria:

1. Known history of traumatic brain injury that required medical care
2. Non-English speaking (based on standardized neuropsychological testing and questionnaires)
3. Claustrophobic, the presence of metallic braces, implants or medical devices that are unsafe at 3T or 7T and/or interfere with the MRI/MRS signals

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Teenagers before 22 at the time of consent diagnosis with a Central Nervous System demyelinating disorder.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
MRI Brain without contrast | 10-14 months
  3T MRI
MRI Brain without contrast | 10-14 months
  7T MRI
Change in Score of Delis-Kaplan Executive Function System (D-KEFS) Color | 10-14 months
  Executive Functioning
Change in Score of Word Interference Test (CWIT) | 10-14 months
  Executive Functioning
Change in Score of Symbol Digit Modalities (SDMT)- Oral Version | 10-14 months
  Processing Speed
Change in Score of Beery-Buktencia Developmental Test of Visual-Motor Integration, Sixth Edition (VMI-6) | 10-14 months
  Visual-Motor Integration
Change in Score of Wechsler Intelligence Scale for Children-5th edition (WISCV) | 10-14 months
  Simple Auditory Attention
Change in Score of Wechsler Adult Intelligence Scale-Fourth edition (WAIS-IV) Digits Forward | 10-14 months
  Simple Auditory Attention
Change in Score of WISC-V or WAIS-IV Digits Backward | 10-14 months
  Working Memory
Change in Score of California Verbal Learning Test- Children's Version (CVLT-C) or California Verbal Learning Test-Second Edition (CVLT-II) | 10-14 months
  Verbal Learning and Memory
Change i Score of D-KEFS Letter and Category Fluency | 10-14 months
  Verbal Fluency
Change in Score of WASI-II | 10-14 months
  Estimate of IQ
Change in Score of Woodcock-Johnson Tests of Achievement Letter Word identification | 10-14 months
  Basic Reading Skill
Change in Score of Reading Fluency | 10-14 months
  Reading Speed
Change in Score of Calculation | 10-14 months
  Math Calculation Skills
Change in Score of Math Fluency | 10-14 months
  Math Speed
Change in Score of Word Attack | 10-14 months
  Phoneme/Grapheme Knowledge
Change in Score of Grooved Pegboard | 10-14 months
  Bilateral Fine Motor Speed and Dexterity
Change in Score of Trail Making Test, Part A and B | 10-14 months
  Simple and complex Attention
Change in Score of Conners Continuous Performance Test 3rd Edition | 10-14 months
  Sustained Attention and Behavioral Inhibition

SECONDARY OUTCOMES:
Change in Examination of Optical Coherence Tomography | 10-14 months
  Eye examination
Change in PROMIS Mobility score | 10-14 months
  Patient Reported Outcomes Measures: Mobility, walking
Change in PROMIS Pain score | 10-14 months
  Patient Reported Outcomes Measures: overall pain level
Change in PROMIS Peer relationship score | 10-14 months
  Patient Reported Outcomes Measures: Peer relationships
Change in PROMIS Stress score | 10-14 months
  Patient Reported Outcomes Measures: Psychological stress
Change in PROMIS Upper extremity movement score | 10-14 months
  Patient Reported Outcomes Measures: Upper extremity movement
Change in score of 25 foot timed walk | 10-14 months
  Walking speed
Change in score of 6 minute timed walk | 10-14 months
  Walking Distance
Change in score of Hauser Ambulation Index | 10-14 months
  Functional walking assessment
Change in score of Multiple Sclerosis Functional Capacity (MSFC) | 10-14 months
  Hand and Eye coordination, Memory test
Change in score of Modified Rankin Scale | 10-14 months
  Disability scale

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Greenberg, MD. MHS, Principal Investigator — University Texas Southwestern
Locations (1):
- University Texas Southwestern, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No